CLINICAL TRIAL: NCT03595826
Title: The Effects of Exercise Therapy on the Co-Morbidity of Attention Deficit and Hyperactivity Disorder (ADHD) and Developmental Co-Ordination Disorder. (DCD)
Brief Title: Co Morbid Attention Deficit and Hyperactivity Disorder(ADHD) and Developmental Co Ordination Disorder (DCD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of KwaZulu (Other)
Responsible Party: Principal Investigator, Pam Dawson, Principal Investigator, University of KwaZulu
Allocation: Non-Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: Co Morbid ADHD and DCD
Record Dates: First submitted 2018-04-22; First posted 2018-07-23 (Actual); Last update posted 2020-11-27 (Actual); Status verified 2020-11

CONDITIONS: Attention Deficit Disorder With Hyperactivity; Developmental Coordination Disorder
Keywords: ADHD/ADD DCD Exercises Neurostimulant Drugs
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Motor Skills Disorders | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: 3 phase quasi experimental design. Diagnosis and intervention.
Who Masked: Investigator
Masking Description: The Pi will not be involved in post intervention testing of the children/participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 1. Neurostimulant pharmaceutical drugs.. (Experimental): 1.Participants receiving medicinal drugs, such as methylphenidate/Ritalin, administered by a medical practitioner, in dosages prescribed by the practitioner, to suit the child.
  Interventions: Drug: Neurostimulant pharmaceutical drugs
- 2. Exercise Intervention (Experimental): Participants receiving a minimum of 8 sessions of exercise intervention, for the duration of an hour each session. Exercises will be to build muscle tone, improve core stability, enhance balance, improve fine and gross motor skills and visual motor integration.
  Interventions: Drug: Neurostimulant pharmaceutical drugs
- 3. Neurostimulants + Exercise intervention (Experimental): See Arms 1 and 2 above. Both interventions administered together: Pharmaceutical drugs plus exercise intervention
  Interventions: Drug: Neurostimulant pharmaceutical drugs
- 4. Control Group (Experimental): Participants will not receive any intervention during the research process. They will be given an intervention after the research is completed.
  Interventions: Drug: Neurostimulant pharmaceutical drugs

INTERVENTIONS:
Drug: Neurostimulant pharmaceutical drugs — The Pi will only administer the exercise intervention. This will consist of minimum of 8 sessions of group exercises, working on improving muscle tone, core stability, balance, fine and gross motor skills and visual motor integration. The pharmacological therapy will be administered and monitored by medical practitioners, as is the norm with most children diagnosed and treated for ADHD/ADD. Parents of participants will remain responsible entirely for the monitoring of the pharmacological therapy of their children.
  Other Names: Exercise intervention; Neurostimulants + Exercise intervention; Control Group

SUMMARY:
This study aims to establish and present the prevalence figures and demographics of the co-morbidity of ADHD and DCD.

It further aims to design an exercise intervention, to be utilised in the management of the symptoms of both conditions.

Furthermore, it aims at establishing the efficacy of this exercise intervention, when compared with the current and most commonly used intervention, that is: neurostimulant drugs.

DETAILED DESCRIPTION:
This study is an experimental design, having three phases. The study looks at children, aged 8 to 9, in remedial units or LSEN classes, in and around Durban, Kzn, SA; who have been diagnosed with ADHD/ADD.

Phase 1: Teachers of the children identified with ADHD/ADD, will be asked to complete a modified teacher Conner's rating, to confirm the diagnosis of ADHD/ADD. The parent will then be asked to complete a DCD questionnaire (DCDQ) to give the PI an idea of whether co-ordination difficulties exist. The PI will then administer a Motor Assessment Battery for Children (MABC) to confirm the diagnosis of DCD. From the scores derived from the 3 above tests, co-morbidity will be diagnosed. The prevalence figures of co-morbidity will be calculated and presented. Demographics of prevalence figures will be given: Gender, Population group, average age.

Phase 2: The exercise intervention will be designed, drawing from the literature and similar interventions already used in various publications.

This programme will be validated by experts (Physiotherapists and O.Ts from special needs schools) and when 70% consensus is reached on all aspects of the programme, the final version will be drafted.

Phase 3: The children found to have both conditions, in co-morbidity, will be assigned to one of 4 groups, according to parental choice, medical advice from paediatricians, GPs etc and an intervention a child is already on.

The four groups will be: medication, exercises, medication plus exercises and a control group. The intervention designed in phase 2 will be administered to the two groups opting for the exercise intervention, for a minimum of 8 sessions. The 3 pre intervention scores (Conner's, DCDQ and MABC) will be derived from phase 1, post intervention scores will be done 6 months after completion of the intervention, as it is stipulated by the rules of the MABC that the test may not be repeated sooner. The pre and post intervention scores will be compared to calculate improvement and average improvement within each group, will be calculated, to establish which intervention or combination of interventions, is the most effective.

ELIGIBILITY:
Inclusion Criteria:

* Age 8 to 9, diagnosed with ADHD, in remedial unit or LSEN class, in mainstream school in Durban Kzn SA.

Exclusion Criteria:

* Any child having an obvious physical disability, neurological condition, musculoskeletal condition, psychiatric disorder or genetic disorder.

Any child below age 8 and above age 9.

Ages: 8 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 151 (Actual)
Dates: Start 2018-05-02 (Actual); Primary Completion 2019-05-30 (Actual); Study Completion 2019-05-30 (Actual)

PRIMARY OUTCOMES:
Inattention, impulsivity and hyperactivity will be rated, using Conners rating scale. | Aproximately 6 months
  Improvement or regression in symptoms of ADHD will be rated using the modified Conner's teacher rating scale, pre intervention and post intervention:
  10 factors on inattention will be rated 0 (Not at all), 1 (Just a little), 2 (Pretty much) and 3 (Very much); 5 factors on impulsivity will be rated using the same scale as above and 5 symptoms of hyperactivity as well. Percentages will be derived from these ratings. A 70% or more indicates a positive diagnosis for inattention/impulsivity/hyperactivity.

SECONDARY OUTCOMES:
Motor co-ordination will be rated, using DCD questionnaire | Aproximately 6 months.
  Improvement or regression in symptoms of co ordination, will be rated by the parent, using the Developmental Co-ordination Disorder Questionnaire, pre and post intervention: 15 statements related to co-ordination will be rated on the following scale: 1 (Not at all like child), 2 (A bit like child), 3 (Moderately like child), 4 (Quite a bit like child) and 5 (Extremely like child). The score will be totalled and scores of 55 and above mean that the child does NOT have co-ordination issues, scores below 55 indicate that the child has co-ordination issues.

OTHER OUTCOMES:
Motor co-ordination will be measured using the Movement Assessment Battery for Children | Aproximately 6 months.
  Improvement or regression of motor/co-ordination symptoms, will be tested by the therapist/primary investigator, using the Movement Assessment Battery for Children. 8 age-appropriate motor tests will be administered and scored.A total Motor Impairment score (TOMI) of under 10,5 indicates that the child is fine, scores from 10,5 to 14 indicate that the child is borderline and scores of 14,5 and above indicate definite motor/co-ordination problems.

CONTACTS AND LOCATIONS:
Overall Officials: Pamela M Dawson, M.Physio, Principal Investigator — Principal Investigator
Locations (1):
- Escombe Primary School, Durban, KwaZulu-Natal, South Africa

IPD SHARING:
Plan to Share IPD: Yes
I plan to share my protocol, study design, intervention, statistical analysis and results. Pretty much the entire study, once comlpeted.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Probably in 2019 and can remain available for as long as is allowed and necessary.
Access Criteria: Clinical trial site.

REFERENCES:
- [Background] Nelson et al. (2015) DCD. Medscape: Drugs, diseases and Procedures.